CLINICAL TRIAL: NCT01498783
Title: Phase I Study of 5-Fluorouracil in Children and Young Adults With Recurrent Ependymoma
Acronym: SJREFU
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJREFU; NCI-2012-00368 (Registry Identifier: NCI Clinical Trial Registratoin Program)
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2015-07

CONDITIONS: Central Nervous System Malignancies; Ependymoma
MeSH Terms: conditions — Ependymoma | interventions — Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Participants meeting the eligibility requirements.
  Intervention: 5-fluorouracil
  Interventions: Drug: 5-fluorouracil

INTERVENTIONS:
Drug: 5-fluorouracil — 5-fluorouracil, bolus dose of 500 mg/m^2 given weekly for 4 weeks followed by a two week rest period equals one cycle (6 weeks). Therapy may continue for up to 16 cycles (about 2 years).
  Other Names: 5-FU

SUMMARY:
This is a phase I study to investigate the safety and pharmacokinetics of weekly 5-fluorouracil (5-FU) administered as a bolus dose in children and young adults with recurrent or refractory ependymoma. The results from this study will inform a subsequent phase II St. Jude investigator-initiated trial.

DETAILED DESCRIPTION:
The initial 5-FU dosage will be 500 mg/m^2 administered on day 1 of course 1. We plan to treat a maximum of 3 cohorts of research participants (dosage levels - 0, 1, and 2) with escalating doses of 5-FU. A cycle is defined as 42 days. The first 6 weeks of therapy will constitute the dose-limiting toxicity (DLT) evaluation period.

Primary objective

* To investigate the safety and pharmacokinetics (plasma and cerebrospinal fluid) of weekly bolus dose 5-FU in children and young adults with recurrent/refractory ependymoma
* To study the safety of 500 mg/m^2 weekly bolus dose 5-FU in less-heavily pre-treated children and young adults with recurrent/refractory ependymoma.

Secondary objectives

* To document and describe toxicities associated with 5-FU administered on a weekly bolus schedule
* To document preliminary antitumor activity in participants with recurrent or refractory ependymoma treated with 5-FU
* To assess the feasibility of measuring expression level of Thymidylate Synthetase (TYMS) in formalin fixed paraffin embedded (FFPE) tumor samples using the Quantigene assay
* To evaluate the association between specific genetic polymorphisms (e.g., DPYD) and the pharmacokinetics of 5-FU

ELIGIBILITY:
INCLUSION CRITERIA:

* Participant must have recurrent or refractory intracranial or spinal ependymoma (including myxopapillary, clear cell, papillary, tanycytic and anaplastic ependymoma or subependymoma). The diagnosis must be confirmed by the pathologist on tissue obtained at either initial diagnosis or at time of recurrence prior to registration.
* Participants may have had two prior systemic anti-cancer chemotherapy regimens, including any chemotherapy, biologic modifiers or small molecules. These may have been given either before or after irradiation.
* Participant must be < 22 years (eligible until 22nd birthday) of age at the time of enrollment.
* Negative testing for DPYD*2 any time prior to enrollment (does not need to be within 7 days)
* Neurologic deficits: Participants with neurological deficits should have a stable or improving neurologic exam for a minimum of 1 week prior to study registration.
* Performance level: Karnofsky Performance Scale (participants > 16 years of age) or Lansky Performance Score (participants ≤ 16 years of age) must be > 30 within two weeks prior to registration.
* Chemotherapy: Participants must have received their last dose of known myelosuppressive anticancer chemotherapy at least four weeks prior to study registration or at least six weeks if nitrosurea. At least two weeks must have lapsed if participants received lower dose oral etoposide (50 mg/m^2) without experiencing evidence of myelosuppression (i.e., neutropenia or requiring transfusion with blood products).
* Biologic agent: Participant must have recovered from any toxicity potentially related to the agent and received their last dose of the biologic agent ≥ 7 days prior to study registration. For biologic agents that have a prolonged half-life, the appropriate interval since last treatment should be discussed with the PI prior to registration.
* Monoclonal antibody treatment: At least three half-lives must have elapsed prior to registration. Such participants should be discussed with the PI prior to registration
* XRT: No more than two prior radiation regimens. For participants who have had prior irradiation for treatment of their ependymoma. XRT must be:

  * ≥ 6 months prior to registration if treated with craniospinal irradiation (≥ 18 Gy)
  * ≥ 4 weeks prior to registration if treated with focal irradiation to the primary tumor
  * ≥ 2 weeks prior to registration if treated with focal irradiation to symptomatic metastatic sites
* Bone marrow or stem cell transplant: Participant must be ≥ 3 months since high dose chemotherapy and peripheral blood stem cell rescue prior to registration
* Anti-convulsants: Participants with seizure disorder may be enrolled if well controlled on anti-epileptic drugs.
* Corticosteroids: Participants who are taking corticosteroids must be on a stable or decreasing dose for at least 1 week prior to registration.
* Growth factors: Participants must be off all colony forming growth factors(s) for at least 1 week prior to registration (e.g. filgrastim, sargramostim, erythropoietin) and at least 2 weeks for long-acting formulations (e.g. Neupogen®).
* Adequate organ function at the time of study enrollment as defined as follows: Laboratory values must be assessed within 7 days prior to registration and must be repeated if initial labs were done greater than 7 calendar days prior to the start of therapy:

  * Bone marrow: Absolute neutrophil count (ANC) ≥ 500/μL, platelet count ≥ 50,000/μL (transfusion independent), hemoglobin concentration ≥ 8g/dL (may be transfused)
  * Renal: Normal serum creatinine concentration based on age or GFR > 70ml/min/1.73m^2
  * Hepatic: Total bilirubin concentration < 1.5x the institutional upper limit of normal for age; SGPT and SGOT < 2.5 x the institutional upper limit of normal

EXCLUSION CRITERIA:

* Participants may not have been previously treated with 5-FU
* Participants receiving any other anticancer or experimental treatment
* Participants with uncontrolled infection
* Participants with any concomitant significant medical illness that in the investigator's opinion cannot be adequately controlled with appropriate therapy, or that would compromise the participant's ability to tolerate therapy, impair the evaluation of side effects related to this treatment, or alter drug metabolism
* Females of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to study entry.
* Participants of child bearing potential must agree to use an effective contraceptive method.
* Participants must not breastfeed while on this study

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2011-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Estimate the maximum tolerated dose determined using the Rolling 6 design using the CTCAEv4 to assess DLT. | At the end of the 6-week dose limiting toxicity observation period.
  To investigate the safety and pharmacokinetics (plasma and cerebrospinal fluid) of weekly bolus dose 5-fluorouracil (5-FU) in children and young adults with recurrent/refractory ependymoma
Pharmacokinetic modeling of 5-fluorouracil concentrations | Pharmacokinetics on day 1, day 8, and day 22 of course 1, and day 1 of course 2
  To investigate the safety and pharmacokinetics (plasma and cerebrospinal fluid) of weekly bolus dose 5-fluorouracil (5-FU) in children and young adults with recurrent/refractory ependymoma
Estimate the maximum tolerated dose in less heavily pre-treated children | At the end of the 6-week dose limiting toxicity observation period.
  To investigate the safety and pharmacokinetics (plasma and cerebrospinal fluid) of weekly bolus dose 5-fluorouracil (5-FU) in children and young adults with recurrent/refractory ependymoma and in less heavily pre-treated children.

SECONDARY OUTCOMES:
Descriptive report of toxicities. | Throughout treatment, up to two years per patient
  To document and describe toxicities associated with 5-FU administered on a weekly bolus schedule
Tumor response and progression-free survival | at the completion of therapy (2 years)
  To document preliminary antitumor activity in participants with recurrent or refractory ependymoma treated with 5-FU
Expression level of TYMS in FFPE tumor samples | At the end of accrual (3 years)
  To assess the feasibility of measuring expression level of Thymidylate Synthetase (TYMS) in formalin fixed paraffin embedded (FFPE) tumor samples using the Quantigene assay
Description of association between genetic polymorphism and pharmacokinetics | At the end of therapy (2 years)
  To evaluate the association between specific genetic polymorphisms (e.g., DPYD) and the pharmacokinetics of 5-FU

CONTACTS AND LOCATIONS:
Overall Officials: Clinton F. Stewart, PharmD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols